CLINICAL TRIAL: NCT02138318
Title: Randomized Controlled Trial of High Definition White Light Endoscopy Versus Chromoendoscopy for Dysplasia Detection in Ulcerative Colitis Surveillance
Brief Title: High Definition Versus Chromoendoscopy for Dysplasia Detection in Ulcerative Colitis (UC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA12/10210
Record Dates: First submitted 2014-04-01; First posted 2014-05-14 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chromoendoscopy (Other)
  Interventions: Other: chromoendoscopy
- High definition (HD) endoscopy (Other)
  Interventions: Other: High definition (HD) endoscopy

INTERVENTIONS:
Other: High definition (HD) endoscopy
  Arms: High definition (HD) endoscopy
Other: chromoendoscopy
  Arms: chromoendoscopy

SUMMARY:
Patients with ulcerative colitis (UC) have an increased risk for colorectal cancer (CRC) compared to the general population. Regular screening by colonoscopy is an internationally recommended cancer prevention strategy. Random sampling of the mucosa throughout the colon has been the mainstay of conventional surveillance practice to detect abnormalities, known as dysplasia which can progress to CRC. This requires multiple biopsies, to be taken and processed, a practice which is is tedious, expensive, time consuming and has a low pickup rate. Dysplasia in UC is typically flat and patchy and can be easily overlooked with standard conventional white light colonoscopy (WLC).

Detection can be improved by the application of dyes which highlight more subtle abnormalities. This practice, known as chromoendoscopy (CE) is better than WLC at dysplasia detection but more time consuming for the patient and cannot guarantee that the whole colon is covered. CE has only been compared in clinical trials with standard definition endoscopy rather than the recently available high definition endoscopes with better resolution and picture. High definition (HD) endoscopy uses a high definition onitor and a high resolution CCD (charge coupled device) providing much better images than standard video endoscopy. HD colonoscopy promises therefore to provide an alternative to CE in UC surveillance without the need for the extra time and experience required for dye spraying for both endoscopists and nursing staff.

The investigators plan to do a randomized trial to assess HD colonoscopy alone compared to chromoendoscopy (with HD colonoscopies) for dysplasia detection during surveillance for ulcerative colitis. There have been no trials comparing these two modalities and the investigators hope to provide evidence that the additional benefit of CE over HD colonoscopy would be marginal and therefore CE would be reserved for procedures using standard definition scopes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with longstanding (more than 10 years), extensive (extending proximal to the splenic flexure) colitis attending for surveillance colonoscopy.
* Patients over 18 years of age

Exclusion Criteria:

* Pregnancy
* Unwilling or unable to give informed consent
* Severe active colitis (as assessed by the endoscopist)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2015-09-19 (Actual); Study Completion 2015-09-19 (Actual)

PRIMARY OUTCOMES:
number of lesions | Once annually at routine clinical assessment
  The number of lesions with at least low grade dysplasia detected by targeted biopsy to be compared between the two groups by chisquared test.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom